CLINICAL TRIAL: NCT06110091
Title: Multi-center Trial to Improve Nocturia and Sleep in Older Adults (MINT)
Brief Title: Multi-center Trial to Improve Nocturia and Sleep in Older Adults
Acronym: MINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Collaborators: VA Greater Los Angeles Healthcare System (U.S. Federal Agency); Emory University (Other); University of California, Los Angeles (Other); University of California, San Francisco (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Elizabeth Camille Vaughan, Principal Investigator, Atlanta VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00006141
Record Dates: First submitted 2023-10-16; First posted 2023-10-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Nocturia; Insomnia
MeSH Terms: conditions — Nocturia; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Behavioral Therapy Program (Experimental): Integrated Behavioral Therapy consists of 5 weekly one-hour sessions (face-to-face either through video or in-person) + 2 telephone check-in with an interventionist. This program integrates cognitive-behavioral treatment for nocturia and insomnia. Brief telephone check-ins will be comprised of review of topics discussed during the sessions.
  Interventions: Behavioral: Integrated Behavioral Therapy Program
- Health Education Program (Placebo Comparator): The Health Education Program consists of 5 weekly one-hour sessions (face-to-face either through video or in-person) + 2 telephone check-in with an interventionist. The program modules focus on brain health and includes topics such physical activity, social engagement, sleep topics (e.g., changes in sleep that occur with aging, effects of poor sleep on health), medications/medical conditions, vision and hearing impairment. Brief telephone check-ins will be comprised of review of health topics discussed during the sessions.
  Interventions: Behavioral: Health Education Program

INTERVENTIONS:
Behavioral: Integrated Behavioral Therapy Program — Integrated Behavioral Therapy is a behavioral program that includes education, lifestyle habits management, cognitive, relaxation, and behavioral conditioning for nocturia and insomnia
  Arms: Integrated Behavioral Therapy Program
Behavioral: Health Education Program — Health Education Program modules focus on brain health and includes topics such physical activity, social engagement, sleep topics (e.g., changes in sleep that occur with aging, effects of poor sleep on health), medications/medical conditions, vision and hearing impairment.
  Arms: Health Education Program

SUMMARY:
The Multi-center Trial to Improve Nocturia and Sleep in Older Adults (MINT) study is a randomized trial to determine and assess the efficacy of integrated treatment of coexisting nocturia and insomnia, as well as explore the effects of this treatment on quality of life.

DETAILED DESCRIPTION:
The Multi-center Trial to Improve Nocturia and Sleep in Older Adults (MINT) study is a randomized trial to determine and assess the efficacy of integrated treatment of coexisting nocturia and insomnia, as well as explore the effects of this treatment on quality of life. While prior research suggests the benefits of multicomponent behavioral treatment, there is an urgent need for treatment strategies that also address concomitant sleep factors, and this study has the potential to provide evidence needed for this shift in the recommended treatment of nocturia among older adults. The study population includes men and women aged 60 years or older who have nocturia at least twice nightly based on the International Consultation on Incontinence Questionnaire Overactive Bladder Module (ICIQ-OAB) questionnaire and insomnia symptoms based on the Insomnia Severity Index. Participants will be identified through 5 sources: 1) Computer-based screening using the Veterans Affairs (VA) Corporate Database Warehouse to screen veterans who live close to the Medical Center, as well as data pulling real Social Security Numbers (SSNs) from VA's Information and Computing Infrastructure (VINCI); 2) a survey mailed once at the end of year 1 to individuals aged > 60 years who have received care at VA Greater Los Angeles (VAGLA) and University of California, Los Angeles (UCLA) sleep center and clinics and Atlanta VA and Emory University sleep center and clinics within the past 6 months; 3) referrals from clinic providers; 4) flyers/advertisements posted in the medical centers; and 5) social media advertisements.

Individuals who meet initial screening criteria will be invited to a face-to-face appointment, where participants will provide written informed consent (either paper or e-consent). At the initial screening appointment, participants will be screened for sleep apnea; have their medical records reviewed; be administered questionnaires; have blood and urine tests; and be provided with a wrist actigraph to wear at home for 1 week, along with a sleep and urinary symptom diary to complete while wearing the actigraph. If eligible, participants will be randomly assigned to either the intervention or the control. Participants assigned to Integrated Behavioral Therapy will receive combined cognitive behavioral therapy for insomnia and nocturia delivered by an interventionist, while those assigned to the Health Education Program will be provided with a health education curriculum delivered by the interventionist. After the final session, participants will have a post-intervention assessment and monthly phone calls until the final assessment 4 months later. The post-intervention assessment and 4-month assessment will include many of the same measures from the screening/baseline visit. Overall, participants in either group will receive 2 baseline/screening visits, 5 weekly one hour sessions either in-person or remotely, one post-intervention session, 3 monthly 15-minute phone calls, and 1 final assessment over the span of approximately 4 months.

Our intended sample size is 96 participants in each group across all sites (total of N=192 randomized participants across all sites; n=96 at Atlanta VA, with n=48 randomized to the Integrated Behavioral Therapy and n=48 randomized to the Health Education Program. The investigators expect to complete 392 baseline assessments (196 per site) to reach our intended sample size.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Average of ≥ 2 episodes per night of nocturia on the International Consultation on Incontinence Questionnaire-Overactive Bladder Module (ICIQ-OAB) questionnaire
* Insomnia Severity Index > 7
* Able to attend weekly study visits

Exclusion Criteria:

* Prior cognitive behavioral therapy for insomnia
* Presence of bipolar disorder
* Significant cognitive impairment as measured by a score < 20 on the Mini-Mental State Exam
* Sleep disturbance better explained by another sleep disorder such as restless legs syndrome, narcolepsy, insufficient sleep syndrome, or circadian rhythm sleep-wake disorders
* Untreated sleep-disordered breathing (respiratory event index ≥ 15 plus • Epworth Sleepiness Scale > 10 or respiratory event index > 30. Note that participants with treated sleep-disordered breathing will not be excluded)
* Current urinary tract infection or hematuria
* Unstable doses or recent changes in bladder medication
* New or recently discontinued insomnia medication within past month
* Previous or current intensive behavioral therapy for insomnia or urinary symptoms,
* Unstable health conditions expected to result in death or hospitalization within 3 months, as assessed by overall study PIs or Site PI.
* Unstable medical conditions that could contribute to nocturia or insomnia such as poorly controlled heart failure as evidenced on physical examination, poorly controlled diabetes mellitus with either hemoglobin A1c of ≥ 9.0, or chronic kidney disease (stage 4 or 5) or a potential to initiate dialysis in 3 months
* Unstable psychiatric conditions (e.g., psychosis, active alcohol/substance abuse based on history and medical records)
* Unstable housing situation
* Evidence of significant urinary retention as measured by a residual bladder volume of ≥ 200 mL by bladder ultrasound with 15 minutes of voiding
* Genitourinary cancer undergoing active treatment
* Pelvic or colon surgery within 6 months of enrollment or onabotulinum toxin therapy for urinary symptoms within 6 months of enrollment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Mean Nocturia Frequency | 4 months
  The primary outcome of nocturia frequency will be measured as the average episodes per night at baseline, 2 months, and 4 months through the International Consultation on Incontinence Questionnaire-Overactive Bladder Module (ICIQ-OAB) questionnaire. An adapted version that asks the participant to record the number of nocturia episodes if the "4+" nocturia option is selected will be used. A linear mixed effects model will be used to evaluate the group difference over time in average nocturia frequency per night.

SECONDARY OUTCOMES:
Self-Reported Insomnia Severity Index | 4 months
  The self-reported Insomnia Severity Index is a 7-item instrument with high internal consistency and validity for measures of fatigue, quality of life, anxiety, and depression. The total score is the sum of all seven items and ranges from 0-28 with higher scores indicating greater insomnia severity. The Insomnia Severity Index can also be used as a change score that measures perceived severity of insomnia symptoms. A 0.5 standardized mean difference between treatment and control is considered the clinical significance threshold for studies of chronic insomnia disorder.
  The Insomnia Severity Index will be modeled similarly with a linear mixed mode. If the distributions of the secondary outcome is skewed and no good transformation is found, the outcome will be categorized into categories based on quantiles or clinically meaningful values and then modeled with generalized linear mixed models using cumulative logit or generalized logit link for multinomial data.
Nocturia-Quality of Life | 4 months
  The Nocturia-Quality of Life (NQOL) questionnaire provides a detailed and robust measure to assess the impact of nocturia on quality of life with particular reference to the effects on persons' lives of nocturia and can be used as an outcome measure to assess impact of different treatment modalities. The NQOL score may be calculated by summing all items, giving a score from 0-58. A greater score indicates a higher impact on QOL.
  The NQOL will be modeled similarly with linear mixed models in their original scale or transformed scale as appropriate. If the distributions of the NQOL scores are skewed and no good transformation is found, the outcomes will be categorized into categories based on quantiles or clinically meaningful values and then modeled with generalized linear mixed models. Similar secondary analyses as those proposed in assessing mean nocturia frequency will be performed on the secondary outcomes NQOL.

CONTACTS AND LOCATIONS:
Overall Officials: E. Camille Vaughan, MD, MS, Principal Investigator — Atlanta VAMC & Emory University
Locations (2):
- United States (2):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Atlanta VAHCS, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Fung C, Bolstad CJ, Huang A, Markland A, Cheng J, Alessi C, Johnson TM 2nd, Bliwise DL, Burgio KL, Martin JL, Schembri M, Der-McLeod E, Sergent T, Vaughan C. Protocol for a multi-site randomized trial testing an integrated behavioral treatment for improving nocturia and insomnia symptoms in older adults (MINT). Res Sq [Preprint]. 2025 Sep 25:rs.3.rs-7330051. doi: 10.21203/rs.3.rs-7330051/v1. PMID 41041560